CLINICAL TRIAL: NCT03366311
Title: TCH-Zhong-Xing-Branch-Emergency-Department
Brief Title: TCHCCT-Zhong-Xing-Emergency-Department-airway
Acronym: TT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Hung,Tzu-Yao, Emergency Medicine Physician, Taipei City Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TCHCCT-ZXER
Record Dates: First submitted 2017-11-27; First posted 2017-12-08 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Airway Complication of Anesthesia; Intubation;Difficult
Keywords: intubation; epiglottis lift; hold high position

STUDY DESIGN:
Intervention Model Description: Prospective randomised crossover manikin study
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- holding position (Active Comparator): different holding position of endotracheal tube
  Interventions: Procedure: holding position
- stylet shapes (Active Comparator): banana shape versus straight-to-cuff shape
  Interventions: Procedure: holding position
- epiglottis lift (Active Comparator): with epiglottis lift or without
  Interventions: Procedure: holding position

INTERVENTIONS:
Procedure: holding position — two types of holding positions plus two types of shapes of stylet, with or without epiglottis lift
  Other Names: shapes of stylet; epiglottis lift

SUMMARY:
To investigate which shapes of stylet, hand techniques and possible condition that improve intubation successful rate and reduce the elapsed intubation time.

DETAILED DESCRIPTION:
Challenging airway is always a big issue in emergency room. However, better hand technique, stylet shapes and conditions affecting intubation successful rate, elapsed duration need further investigations. We compare two endotracheal tube holding position, two holding places, with or without epiglottis lift technique in this study. All intubation processes in the study will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* care givers with sufficient understanding of airway anatomy and management

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
intubation successful rate | through study completion, and average of 15minutes
  intubation more than 90 seconds considered as a failed intubation

SECONDARY OUTCOMES:
intubation elapsed time | through study completion, and average of 15minutes
  from insertion of endotracheal to the tube until proper placement of endotracheal tube
insertion elapsed time | through study completion, and average of 15minutes
  from proper glottic view to the tube until proper placement of endotracheal tube
difficulty of intubation | through study completion, and average of 15minutes
  Visual Analogue Scale with a 10cm bar

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Yao Hung, MD, Study Director — Taipei City Hospital ZhongXing Branch
Locations (1):
- Taipei City Hospital Zhong-Xing branch, Taipei, Taiwan

REFERENCES:
- [Derived] Hung TY, Lin LW, Yeh YH, Su YC, Lin CH, Yang TF. The evaluation of a better intubation strategy when only the epiglottis is visible: a randomized, cross-over mannequin study. BMC Anesthesiol. 2019 Jan 10;19(1):8. doi: 10.1186/s12871-018-0663-9. PMID 30630425